CLINICAL TRIAL: NCT02281695
Title: The Influence of Different PEEP Values on Gas Exchange in Spontaneously Breathing Patients During Early Weaning
Brief Title: PEEP Influence on Gas Exchange During Early Weaning
Acronym: MHOPEEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of Primary investigators
Sponsor: Marienhospital Osnabrück (Other)
Responsible Party: Principal Investigator, Studienarzt K2A, P.D. dr. med. Martin Beiderlinden, Marienhospital Osnabrück
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MHO 001
Record Dates: First submitted 2014-10-29; First posted 2014-11-03 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): Patients that are mechanically ventilated for less than 24 hours until the weaning process can be started.
  At the beginning of the weaning process the PEEP will be adjusted at a value equal with the PEEP during BiPAP (Group 1) and Pmean during BiPAP (Group 2) During controlled mechanical ventilation all patients will be for 5 minutes with FiO2 - 100% ventilated. The PaO2/FiO2 after 5 minutes ventilation with 100% oxygen will be compared with the PaO2/FiO2 during ventilation with 30% oxygen.
  Interventions: Other: PEEP adjusment during the Weaning process
- Arm B (Active Comparator): Patients that are mechanically ventilated for more than 24 hours until the weaning process can be started. At the beginning of the weaning process the PEEP will be adjusted at a value equal with the PEEP during BiPAP (Group 1) and Pmean during BiPAP (Group 2) During controlled mechanical ventilation all patients will be for 5 minutes with FiO2 - 100% ventilated. The PaO2/FiO2 after 5 minutes ventilation with 100% oxygen will be compared with the PaO2/FiO2 during ventilation with 30% oxygen.
  Interventions: Other: PEEP adjusment during the Weaning process

INTERVENTIONS:
Other: PEEP adjusment during the Weaning process — The PEEP will be adjusted after an previously established algorithm and the differences in the arterial blood oxygen partial pressure will be compared.

SUMMARY:
The purpose of this study is to determine the differences in oxygenation and decarboxylation between two weaning processes.

DETAILED DESCRIPTION:
First, during controlled mechanical ventilation all patients will be ventilated for 5 minutes with 100% oxygen. After 5 minutes an PaO2/FiO2 will be calculated and compared with a PaO2/FiO2 during ventilation with FiO2 - 30%.

The patients will be divided in two sections: Section A are the patients with less than 24 hours mechanical ventilation until weaning start. Section B are the patients with more than 24 hours until weaning start.

The patients in every section will be further divided in two groups. Group 1 will be weaned starting with a PEEP equal with P mean during BiPAP, Group 2 will be weaned starting with a PEEP equal with PEEP during BiPAP.

Further, the weaning will be conducted after an known algorithm. The differences in the oxygenation and decarboxylation will be measured after 30 and 120 Minutes for Group A and after 30, 120, 240, 360 Minutes for Group B.

ELIGIBILITY:
Inclusion Criteria:

* All Patients that are mechanical ventilated on the intensive care unit.

Exclusion Criteria:

* Patients under 18 years of age
* Patients that where in an other study in the last 30 days
* Patients that are enrolled in other studies
* Pregnant woman
* Nursing mothers
* Existing severe Lung disease
* Existing COPD Gold IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in the Oxygen Partial Pressure and CO2 Partial Pressure in the arterial blood gas analysis | 30, 60, 90, 120, 360 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Martin Beiderlinden, P.D. dr. - med., Principal Investigator — Marienhospital Osnabrück
Locations (1):
- Marienhospital Osnabrück, Osnabrück, Lower Saxony, Germany